CLINICAL TRIAL: NCT05058365
Title: Effects of Mindfulness Training on the Psychological Well-being of Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Lam Shui-fong, Director, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UHongKong(JC PandA)
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Mindfulness-based Intervention for Preschoolers
Keywords: mindfulness, psychological well-being of preschoolers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: dots Curriculum
- Wait-list control (No Intervention): Participants in wait-list control group will receive the same intervention, two months after their counterparts in experimental group completed the intervention.

INTERVENTIONS:
Behavioral: dots Curriculum — dots is a mindfulness curriculum developed by Mindfulness in Schools Project (MiSP) for children aged 3-6 in pre-school settings. The program consists of 15-minute twice weekly lessons that span for fifteen weeks. dots has various suggestions for "Have A Go" after each session - both in the classroom and at home.
  Arms: Intervention group

SUMMARY:
The present study is a randomized controlled trial to evaluate the effectiveness of a mindfulness course on the psychological well-being of preschoolers (i.e., attention and impulsivity, prosocial behavior, empathy, emotion regulation and conduct). Participants will be randomized to either intervention (dots Curriculum) or wait-list control condition. Participants will complete a computerized task and they will be interviewed to complete a scenario test before (baseline) and after the intervention. The parents and class teacher will also be invited to complete a survey at baseline and after the intervention.

ELIGIBILITY:
* Aged 3-6 years
* Studying in pre-school settings

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shui-fong Lam, Principal Investigator — The University of Hong Kong
Locations (1):
- Jockey Club "Peace and Awareness" Mindfulness Culture in Schools Initiative, Faculty of Social Sciences, The University of Hong Kong, Hong Kong, Hong Kong

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A whole grade of K3 kindergarteners was recruited from a kindergarten in Hong Kong.
Period: Overall Study
Arm/Group | Intervention Group | Wait-list Control
Started | 9 | 9
Completed | 8 | 8
Not Completed | 1 | 1
Not completed — Migration | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Wait-list Control | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.556 (0.527) | 5.000000 (0) | 4.778 (0.428)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 9 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Attention and Impulsivity
Description: An aggregated T-score by taking the mean of the eight measures of Conners Kiddie Continuous Performance Test 2nd Edition (K-CPT 2), published by Multi-Health Systems. The eight measures are d-prime, Omissions, Commissions, Perseverations, Hit Reaction Time Standard Deviation, Variability, Hit Reaction Time Block Change, Hit Reaction Time Inter-Stimulus Interval Change. All eight measures were T-score with a population mean of 50 with a standard deviation of 10. The eight T-scores are averaged to give an overall representation of the children's attention and impulsivity. Lower score indicates better outcome.
Time Frame: Baseline, Immediately after intervention at Week 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 8 | 8
units on a scale
  Baseline | 50.05 (8.47) | 53.45 (7.70)
  After training | 48.32 (7.43) | 56.17 (9.31)

2. Primary Outcome: Empathy
Description: Scenario test depicting common social interactions faced by preschoolers. Two parallel versions are developed, each with four scenarios. For each scenario, the children are asked to identify the emotions of the character in the scenario. Answers of the same emotional valence (i.e. positive or negative) without probe score 2 points. Answer after probe score 1 point. Answers with different emotional valence or null responses score 0 points. The mean score of the four scenarios is calculated as the measure of empathy, ranging from 0 to 2. Higher scores indicate stronger empathy.
Time Frame: Baseline, Immediately after intervention at Week 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 8 | 8
units on a scale
  Baseline | 1.53 (0.36) | 1.47 (0.91)
  After training | 1.41 (0.44) | 1.59 (0.67)

3. Primary Outcome: Prosocial Behavior
Description: Scenario test depicting common social interactions faced by preschoolers. Two parallel versions are developed, each with four scenarios. For each scenario, the children are asked to identify the emotions of the character in the scenario. Answers of socially appropriate behaviors without probe score 2 points. Answer of socially appropriate behaviors after probe score 1 point. Answers with socially inappropriate behavior or null responses score 0 points. The mean score of the four scenarios is calculated as the measure of prosocial behavior, ranging from 0 to 2. Higher scores indicate more prosocial behavior.
Time Frame: Baseline, Immediately after intervention at Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 1.38 (0.92) | 1.75 (0.71)
  After training | 1.50 (0.76) | 1.50 (0.76)

4. Primary Outcome: Parent-reported Attention
Description: The mean subscale score of a modified version of the Hyperactivity subscale of the parent-reported Strengths and Difficulties Questionnaire (SDQ). Originally negative Items were changed into positive wording. The subscale consisted of 3 items, rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). Higher score indicated better attention.
Time Frame: Baseline, Immediately after intervention at Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 3.58 (0.43) | 3.46 (0.62)
  After training | 3.54 (0.71) | 3.50 (0.59)

5. Primary Outcome: Parent-reported Emotion Regulation
Description: The mean subscale score of a modified version of the Emotional Problem subscale of the parent-reported Strengths and Difficulties Questionnaire (SDQ). Originally negative Items were changed into positive wording. The subscale consisted of 3 items, rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). Higher score indicated better emotion regulation.
Time Frame: Baseline, Immediately after intervention at Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 3.88 (0.40) | 3.81 (0.55)
  After training | 3.88 (0.43) | 3.88 (0.43)

6. Primary Outcome: Parent-reported Prosocial Behavior
Description: The mean subscale score of a modified version of the Prosocial subscale of the parent-reported Strengths and Difficulties Questionnaire (SDQ). Originally negative Items were changed into positive wording. The subscale consisted of 3 items, rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). Higher score indicated more prosocial behavior.
Time Frame: Baseline, Immediately after intervention at Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 3.67 (0.36) | 4.08 (0.43)
  After training | 4.00 (0.36) | 4.04 (0.52)

7. Primary Outcome: Parent-reported Conduct
Description: The mean subscale score of a modified version of the Conduct Problem subscale of the parent-reported Strengths and Difficulties Questionnaire (SDQ). Originally negative Items were changed into positive wording. The subscale consisted of 3 items, rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). Higher score indicated less conduct problem.
Time Frame: baseline, immediately after intervention at Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 3.42 (0.50) | 3.63 (0.63)
  After training | 3.58 (0.61) | 3.54 (0.35)

8. Primary Outcome: Teacher-reported Attention
Description: The mean subscale score of a modified version of the Hyperactivity subscale of the teacher-reported Strengths and Difficulties Questionnaire (SDQ). Originally negative Items were changed into positive wording. The subscale consisted of 3 items, rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). Higher score indicated better attention.
Time Frame: Baseline, Immediately after intervention at Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 4.17 (0.61) | 3.83 (0.99)
  After training | 4.63 (0.28) | 4.13 (0.56)

9. Primary Outcome: Teacher-reported Emotion Regulation
Description: The mean subscale score of a modified version of the Emotional Problem subscale of the teacher-reported Strengths and Difficulties Questionnaire (SDQ). Originally negative Items were changed into positive wording. The subscale consisted of 3 items, rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). Higher score indicated better emotion regulation.
Time Frame: baseline, immediately after intervention at Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 4.71 (0.45) | 4.33 (0.87)
  After training | 4.96 (0.12) | 4.79 (0.31)

10. Primary Outcome: Teacher-reported Prosocial Behavior
Description: The mean subscale score of a modified version of the Prosocial subscale of the teacher-reported Strengths and Difficulties Questionnaire (SDQ). Originally negative Items were changed into positive wording. The subscale consisted of 3 items, rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). Higher score indicated more prosocial behavior.
Time Frame: baseline, immediately after intervention at Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 3.79 (0.36) | 4.08 (0.43)
  After training | 4.00 (0.36) | 4.04 (0.52)

11. Primary Outcome: Teacher-reported Conduct
Description: The mean subscale score of a modified version of the Conduct Problem subscale of the teacher-reported Strengths and Difficulties Questionnaire (SDQ). Originally negative Items were changed into positive wording. The subscale consisted of 3 items, rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). Higher score indicated less conduct problem.
Time Frame: baseline, immediately after intervention at Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 4.71 (0.28) | 4.42 (0.66)
  Weew | 4.96 (0.12) | 4.46 (0.47)

ADVERSE EVENTS:
Time Frame: 99 days (the duration of the training period)
Arm/Group | Intervention Group | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT05058365/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT05058365/ICF_001.pdf